CLINICAL TRIAL: NCT01722916
Title: Pilot Study of Appropriate Dosing for Reducing and Removing Hyaluronic Acid Filler With Hyaluronidase: A Randomized Control Clinical Trial
Brief Title: Reducing and Removing Hyaluronic Acid Filler With Hyaluronidase
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery and Surgery-Organ Transplantation, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU68166
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Drug Safety
MeSH Terms: interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose of Hyaluronidase (Experimental)
  Interventions: Drug: Hyaluronidase

INTERVENTIONS:
Drug: Hyaluronidase

SUMMARY:
The purpose of this study is to find how much hyaluronidase should be used when receiving injections of fillers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* The subjects are in good health
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator

Exclusion Criteria:

* Under 18 years of age
* Pregnancy or Lactation
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness
* Recent Accutane use in the past 6 months
* Subjects prone to hypertrophic and keloidal scarring
* Subjects with tattoos and/or scars on upper medial arms (the treatment area)
* Subjects with known hypersensitivity to hyaluronic acid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2012-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose of hyaluronidase injected until the filler is no longer detectable | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Alam M, Hughart R, Geisler A, Paghdal K, Maisel A, Weil A, West DP, Veledar E, Poon E. Effectiveness of Low Doses of Hyaluronidase to Remove Hyaluronic Acid Filler Nodules: A Randomized Clinical Trial. JAMA Dermatol. 2018 Jul 1;154(7):765-772. doi: 10.1001/jamadermatol.2018.0515. PMID 29710212